CLINICAL TRIAL: NCT07376993
Title: Pulse Signal Acquisition in Patients With Heart Failure
Acronym: TCM PA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Temasek Polytechnic, Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-2338; MOE-MOE2020-TIF-0005 (Other Grant/Funding Number: MOE TRANSLATIONAL R&D AND INNOVATION FUND (TIF))
Record Dates: First submitted 2025-07-01; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Pulse signal measurement using measurement device
  Interventions: Device: Pulse Measurement

INTERVENTIONS:
Device: Pulse Measurement — TCM pulse signal data will be collected using project group developed pulse data collector, the collected TCM pulse signal is visible on the collector display screen. Project staff will place the pulse collector cuff on the wrist of the participant. During the process, the airbag in the cuff will be inflated with air several times to press the pressure sensor against participants' wrist and deflated several times to release the pressure. Under different airbag pressure, the TCM pulse signal from different depths (Fu, Zhong, and Chen) against the wrist will be collected. During the test, the project staff will move the cuff along the wrist to collect the TCM pulse signal from different wrist positions (Cun, Guan, and Chi) according to TCM theory.

SUMMARY:
Heart Failure (HF) is usually a chronic condition that gradually gets worse. The heart muscle becomes weaker and has trouble pumping blood to nourish the cells in human body. General symptoms are breathlessness, fatigue, ankle swelling. Accurate and timely diagnosis is crucial to ensure patients receive appropriate treatment. Patients often present to primary care clinicians, however diagnosis by primary care clinicians is inaccurate as symptoms and signs commonly overlap with other conditions. Only 26% of patients with a suspected HF have a confirmed diagnosis after formal investigation according to diagnostic criteria. There is a strong demand to develop an accurate, easy-to-use, costeffective device to detect HF in primary clinics or even by patients themselves before it is too late to modify the natural history of the disease.

TCM palpation provides a simple, cheap, and non-invasive approach for diagnosis and evaluation of the severity of HF, and does not involve use of expensive equipment. There are several specific pulse patterns associated with the clinical manifestation of HF. One of the project collaborators, a TCM physician with a PhD in Chinese Medicine, explained that patients with HF usually have alternating pulse strengths, strong pulse and subsequent weak pulses. The various degrees of severity can be readily manifested as Jiemai, Cumai, and Daimai on the pulse palpation. Based on the investigators' preliminary sensor test results, these pulse features can be easily detected using a micro tubular epidermal sensor, likewise developed by the investigators. Therefore, the investigators propose to use their micro tubular epidermal sensor to develop a TCM pulse analyser, which can be used by primary care clinicians and patient themselves to detect HF in a timely and accurate manner.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 years and above.
* The recruited patients should have been diagnosed by NHCS's Doctor in charge with HF.
* Ability to provide informed consent.

Exclusion Criteria:

- Pregnant Women as their TCM pulse signal maybe different from normal (non-pregnant) time.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
AI-developed Heart Failure detection algorithm | On the day of enrollment
  To develop pulse pattern feature extraction, selection, and classification models using AI approaches with a premier focus on HF detection, based on TCM theory.
Pulse data acquisition from HF patients and non-HF people | On the day of enrollment
  To collect pulse data from HF patients and non-HF people to train and test the machine learning models developed based on AI methods.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided